CLINICAL TRIAL: NCT06645691
Title: Hyperpolarized MR Imaging with Carbon-13 Pyruvate in the Human Body
Acronym: POLARIC-13
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart Centre Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: POLARIC-13
Record Dates: First submitted 2024-10-02; First posted 2024-10-17 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure; Cardiometabolic Syndrome; Cancer Diagnosis; Cardiovascular Diseases; Healthy Volunteers
Keywords: Carbon-13 Pyruvate; Magnetic Resonance Imaging; Lactate; Alanine; Bicarbonate; Hyperpolarized Pyruvate (13C) Injection
MeSH Terms: conditions — Heart Failure; Metabolic Syndrome; Cardiovascular Diseases | interventions — Pyruvic Acid

STUDY DESIGN:
Intervention Model Description: This is a cross-sectional study conducted in healthy volunteers and patients with cardiovascular/cardiometabolic diseases.
  Hyperpolarized 13C-pyruvate will be injected intravenously to participants and the metabolized products will be imaged in real time using MRI scanner. The goal is to determine normal values of glucose metabolism in healthy volunteers and study the potential applications of hyperpolarized imaging in patients with cardiovascular/cardiometabolic diseases.
  All patients will be invited to participate in a repeat scan with the same imaging protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hyperpolarized Pyruvate [13C] Injection (Experimental): Hyperpolarized 13C-pyruvate is injected intravenously at a dose of 0.43 mL/kg body weight, and at a rate of 5 mL/second followed by a 20 mL saline flush at 5 mL/second when the patient is already in the MRI scanner.
  Interventions: Drug: Hyperpolarized 13C-pyruvate

INTERVENTIONS:
Drug: Hyperpolarized 13C-pyruvate — Hyperpolarized 13C-pyruvate is injected intravenously at a dose of 0.43 mL/kg body weight, and at a rate of 5 mL/second followed by a 20 mL saline flush at 5 mL/second when the patient is already in the MRI scanner
  Other Names: (13C) pyruvate; Hyperpolarized Carbon C 13 Pyruvate

SUMMARY:
Positron emission tomography with 18F fluorodeoxyglucose (FDG) is the conventional imaging technique to provide information regarding tissue glucose uptake and has been highly clinically successful. However, it cannot assess downstream metabolism, which may be useful in the diagnosis and assessment of treatment response in a variety of diseases. Patients will also be exposed to ionizing radiation, the amount of exposure can vary depending on the dose of tracer administered, frequency of scans and duration of each scan. Carbon-13 (13C) magnetic resonance imaging (MRI) is particularly attractive for metabolic imaging because carbon serves as the backbone of nearly all organic molecules in the body. With this technique, the polarization increases to approximately 30%-40%, an increase of over 10,000 to 100,000-fold, thereby dramatically increasing the MRI signal . Whilst the role of 13C imaging has been demonstrated in many sites around the world, we aim to demonstrate the feasibility and application of 13C hyperpolarized imaging in healthy Singapore residents and patients with cardiovascular and/or cardiometabolic diseases.

DETAILED DESCRIPTION:
Positron emission tomography with 18F fluorodeoxyglucose (FDG) is the conventional imaging technique to provide information regarding tissue glucose uptake and has been highly clinically successful. However, it cannot assess downstream metabolism, which may be useful in the diagnosis and assessment of treatment response in a variety of diseases. Patients will also be exposed to ionizing radiation, the amount of exposure can vary depending on the dose of tracer administered, frequency of scans and duration of each scan.

Carbon 13 (13C) magnetic resonance imaging (MRI) is particularly attractive for metabolic imaging because carbon serves as the backbone of nearly all organic molecules in the body. However, the low natural abundance of the 13C isotope at ~1.1% has made in vivo imaging extremely challenging. To improve the MR signal 13C nuclei, probes are synthetically enriched to increase the concentration of the 13C label in a molecule. MRI signal can be further increased by the process of hyperpolarization. At low temperature and high magnetic field, electrons have a very high level of polarization (ie, nearly all the electrons are aligned in the same direction). This high level of polarization can be transferred to 13C-labeled probes, increasing their MRI signals. This transfer of polarization is accomplished by mixing radicals (a source of free electrons) with the 13C-labeled probe(s) to be hyperpolarized and placing the mixture in a polarizer at a magnetic field typically of 3.0-5.0 T and at a low temperature (approximately 1 K). Microwave irradiation is then applied to transfer the polarization from unpaired electrons in a trityl radical to the 13C-labeled probe. The final solution retains a high level of polarization and can be formulated to be at physiologic pH, osmolarity, and temperature for in vivo injection and metabolic investigations.

With this technique, the polarization increases to approximately 30%-40%, an increase of over 10,000 to 100,000-fold, thereby dramatically increasing the MRI signal (Figure 1). The enhanced signal, however, is typically available only for a short period of time (1-2 minutes), as the polarization decays back to its thermal equilibrium level. Therefore, rapid imaging is needed to acquire high signal-to-noise ratio metabolic data with minimal polarization loss and to measure fast metabolic processes.

To date, hyperpolarized imaging technique has been performed in more than 800 healthy volunteers and patients; and in more than 1,200 studies in various clinical conditions.

HYPOTHESIS AND OBJECTIVES:

This proof-of-concept study to demonstrate feasibility and application of 13C hyperpolarized imaging in healthy Singapore residents and patients with cardiovascular/cardiometabolic diseases.

1. To establish reference ranges in the metabolic products of hyperpolarized 13C-pyruvate (lactate, alanine and bicarbonate) in healthy volunteers and examine repeatability of the 13C hyperpolarized imaging sequences.
2. To develop the application of 13C hyperpolarized imaging in patients with cardiovascular and cardiometabolic diseases.

ELIGIBILITY:
Inclusion Criteria:

Healthy Volunteers:

1. Age 21 years and above
2. No significant medical co-morbidities (such as chronic kidney disease, diabetes mellitus, heart failure, ischemic heart disease, previous strokes)
3. No history of cancer
4. Able and willing to comply with study procedures and provide signed informed consent

Patients with cardiovascular/cardiometabolic diseases:

1. Age 21 years and above
2. Physician diagnosed cardiovascular conditions: ischemic heart disease, inherited cardiomyopathies (hypertrophic, dilated or infiltrative cardiomyopathies) and stable heart failure; and/or
3. Cardiometabolic conditions (such as diabetes on medications, hypertension, central obesity, fatty liver disease)
4. Able and willing to comply with study procedures and provide signed informed consent

Exclusion Criteria:

1. Standard contraindications for magnetic resonance procedures (such as implantable medical devices, suspected presence of surgical apparatus or shrapnel, severe claustrophobia)
2. Unstable medical conditions (such as symptomatic heart failure, unstable hypertension/glucose levels as determined by investigators, symptomatic arrhythmias, angina)
3. Pregnant or nursing women
4. Known allergies to pyruvate or any of its components

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility and reproducibility of Imaging Technique | 30 - 45 minutes post dose
  Feasibility and reproducibility of the imaging technique in healthy volunteers and patients with cardiovascular and/or cardiometabolic diseases

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No